CLINICAL TRIAL: NCT06934278
Title: Pooled Human Plasma vs Crystalloid in The Management of Children Undergoing Instrumented Spinal Fusion for Scoliosis: A Double-Blind, Randomized Clinical Trial
Brief Title: Pooled Human Plasma vs Crystalloid in The Management of Children Undergoing Instrumented Spinal Fusion for Scoliosis
Acronym: OCTAGON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T/210/2024
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Neuromuscular Scoliosis
Keywords: adolescent idiopathic scoliosis; neuromuscular scoliosis; pooled human plasma; randomized clinical trial; double-blind placebo controlled

STUDY DESIGN:
Intervention Model Description: A double-blind placebo controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pooled human plasma (Active Comparator): Pooled human plasma (Octaplas, 10mL/kg, max 400 mL)
  Interventions: Drug: Pooled human plasma
- Placebo (Placebo Comparator): Crystalloid infusion (Plasmalyte, 10 mL/kg, max 400 mL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pooled human plasma — Infusion of pooled human plasma (Octaplas, 10 mL/kg, max 400 mL) over 1 hour after induction of general anaesthesia
  Arms: Pooled human plasma
Drug: Placebo — Infusion of cryst (Octaplas, 10 mL/kg, max 400 mL) over 1 hour after induction of general anaesthesia
  Arms: Placebo

SUMMARY:
OCTAGON trial is a randomized, double-blinded, parallel-group non-inferiority multicenter (Helsinki and Turku University Hospitals, Finland) clinical trial according to CONSORT criteria.

194 adolescents with idiopathic (major curve > 45 degrees) or neuromuscular scoliosis (major curve > 50 degrees) are enrolled for the OCTAGON trial comparing pooled human plasma (Octaplas, 10mL/kg, active management) vs. Plasmalyte (10 mL/kg, placebo) before incision as part of the normal intraoperative fluid therapy. Data is collected at baseline and at each follow-up until a minimum of 2-year follow-up.

Outcomes Outcomes for the OCTAGON trial include 1) intraoperative blood loss (in mL, primary outcome) and the need for allogenic red blood cell infusion (percentage of patients). Secondary outcomes include health-related quality of life (Scoliosis Research Society 24 outcome questionnaire), postoperative pain (48-hour opioid consumption), operative time (hours), drain output (mL), hidden blood loss (mL), hospital stay, and complications (skin reactions, TRALI, deep surgical site infection, neurologic deficit).

Research questions and hypothesis Does prophylactic use of pooled human plasma decrease intraoperative blood loss in adolescents undergoing instrumented spinal fusion for scoliosis? We hypothesize that pooled human plasma will reduce intraoperative and total blood loss by 25% resulting in lower need for blood transfusion and fewer surgical site infections.

Objectives To compare the effect of pooled human plasma vs. crystalloid fluids on intraoperative bleeding and total blood loss (drain output and hidden blood loss) in children undergoing posterior spinal fusion for AIS and NMS. Adverse events will be recorded and reported as minor (skin reaction) or major (severe allergic reaction, transfusion related acute lung injury, TRALI, deep surgical site infection, neurologic injury).

Ethical aspects The PHP trial has been evaluated via European regulatory authority (EU CT: 2024-514857-31-00) and by Fimea (FIMEA/2024/006588). Informed consent is obtained from the parent(s). Results will be disseminated in high-quality peer-reviewed publications.

The individual patient safety and high-quality management of fractures and scoliosis is a priority in this trial. The randomization can be opened at any stage of the treatment process. Based on the clinical decision the randomized treatment can be terminated and treatment provided accord-ing to clinical decision making even if results will be evaluated using the intention to treat princi-ple. Pain management will be prioritized in every clinical scenario and parental presence is always possible.

DETAILED DESCRIPTION:
Introduction Total blood loss including intraoperative, drain output, and hidden blood loss equals to 40% of blood volume in patients undergoing posterior spinal fusion for paediatric spinal deformities. Despite the perioperative use of tranexamic acid and gelatine matrix with human thrombin, 14% of patients with adolescent idiopathic scoliosis (AIS) and 73% of patients with neuromuscular scoliosis (NMS) require allogenic red blood cell infusion (Soini et al. NASSJ 2022). Early use of pooled human plasma (PHP) may reduce total blood loss in these patients, but there are no studies in the paediatric population undergoing major surgery on this subject.

Objective To compare pooled human plasma (PHP, OCTAPLAS) vs. crystalloid (PLASMALYTE, comparator) for intraoperative bleeding, drain output, and hidden blood loss as well as the sum of these components (total blood loss) in children undergoing posterior spinal fusion for AIS. Adverse events will be recorded and reported as minor (skin reaction) or major (severe allergic reaction, transfusion related acute lung injury, TRALI; deep surgical site infection, neurologic injury). The investigators hypothesize that the use of PHP in the early perioperative management will reduce intraoperative blood loss (primary outcome), drain output, and hidden blood loss accounting for total blood loss and reduce the need for perioperative allogenic red blood cell infusion (secondary outcome) without increasing the risk for adverse events. Additionally, postoperative pain (opioid consumption and pain score, secondary outcome) may be decreased.

Outcomes Primary outcome is intraoperative blood loss (blood loss in mL after wound closure). Secondary outcomes include need for allogenic red blood cell infusion (percentage of patients at hospital release, health-related quality of life (Scoliosis Research Society 24 outcome questionnaire), postoperative pain (48-hour opioid consumption, pain visual analogue score), operative time (hours), drain output (mL), hidden blood loss (mL), hospital stay, and complications (skin reactions, TRALI, deep surgical site infection). Disease specific Scoliosis Research Society (SRS)-24 questionnaires are filled out preoperatively, at 6 months and 24 months during postoperative outpatient clinic visits.

Study design A randomized, double-blinded, multicenter (Helsinki and Turku University Hospitals, Finland) clinical trial according to CONSORT criteria.

After randomization, patients will be given in a blinded fashion (except for anaesthesia nurse) either 10 ml/kg (maximal dose 400 ml) pooled human plasma (OCTAPLAS or 10ml/kg (maximal dose 400 ml) crystalloid (PLASMALYTE) as an intravenous 1-hour infusion, as part of the standard anaesthesia of scoliosis surgery, starting at one hour before incision.

Scoliosis surgery is a complex procedure, in addition to standard pharmacological treatment and anaesthesiologic control of blood pressure, surgical technique significantly affects blood loss during surgery. To dependently determine the effectiveness of OCTAPLAS to reduce blood loss, the operating room needs to be blinded for intervention.

Selection of study population Trial subjects consist of individuals who are planned to undergo PSF for scoliosis as standard practice. Individuals are 10 to 21 years of age. The study population consists of adolescents with idiopathic scoliosis (over 45 degrees) and neuromuscular scoliosis (over 50 degrees).

All individuals are required to give informed consent either by patient, legal representative/parent, or both, when appropriate. Patients under legal age of independent consent (less than 15 or 18) need parents' or caretakers' consent in addition to their own consent. Some neuromuscular scoliosis patients are not capable of giving their own informed consent. In that case the consent is given only by the child´s legal representative or parent.

Suitability for this trial is determined by the need of surgical intervention for scoliosis, thus the patient population who would benefit from the treatment under investigation includes individuals who are minors or are not capable of giving informed consent, thus inclusion of this patient population in this investigation is justified. The clinical trial is essential with respect to incapacitated subjects and data of comparable validity cannot be obtained in clinical trials on persons able to give informed consent, or by other research methods, and the incapacitated subjects have received the information referred to in Article 29(2) in a way that is adequate in view of their capacity to understand.

The sponsor considers that the conditions for the inclusion of incapacitated subjects in the trial, as laid out in Art 31 of the CTR, are considered fulfilled.

Inclusion criteria Subjects meeting all the criteria below may be included in the study. To be eligible for inclusion, each subject must meet each of the following criteria at Screening and must continue to fulfil these criteria at Baseline (Visit 1).

Patients will be included in the study if they fulfil the following criteria:

* Written informed consent.
* Aged between 10 and 21 years of age
* Scoliosis requiring posterior scoliosis surgery using all pedicle screw technique for AIS (>45-degree major curve) or NMS (>50-degree major curve);
* Normal whole spine MRI except for the spinal deformity (only for patients with adolescent idiopathic scoliosis as patients with neuromuscular scoliosis do not typically undergo MR images as they would need general anaesthesia).

Exclusion criteria

Subjects are excluded from the study if any of the following criteria is met at Screening or at Baseline:

* Immunoglobulin A-deficiency
* Need for anteroposterior surgery
* Need for three column vertebral resection
* Smoking
* Diabetes mellitus
* Abnormalities in blood coagulation (thromboplastin time below above or below of normal values, 70-130%)
* Blood trombosytes less than 150 x E9/l
* Body mass index over 40
* Allergy or hypersensitivity to study medications or their ingredients
* Pregnancy or breast-feeding, aim of becoming pregnant during the study.
* Participation in another study and receipt of any other investigational agent during 2 year period of current investigation
* Inability to provide written informed consent
* Any significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk by participation in the study, or may influence the result of the study.
* A history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Known history of, or documented positive hepatitis B or C or HIV infection
* Prior or concurrent malignancy 12
* Aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 3 x upper-limit of normal
* Creatinine clearance (CrCl) < 60 ml/min measured by 24-hour urine collection or estimated from the Cockcroft and Gault formula
* Clinically significant ECG findings as judged by the investigator
* Amiodarone medication
* Hyperkalemia
* Renal insufficiency
* AV-block
* Metabolic or respiratory alkalosis
* Hypochlorhydria
* Hypersensitivity for active component or additives
* Contraception requirements:

Combined hormonal contraception should be stopped 4 weeks prior to receiving IMP. Progestin-only contraceptives including pills, implant and intrauterine system, and Copper IUD) and sexual abstinence are allowed forms of contraception.

Withdrawal Patient can withdraw from trial at any point at will. The infusion is administered during anesthesia and primary outcome can be evaluated in all patients.

Randomization and blinding The randomization is carried out by research coordinator, using a computer-generated method (www.sealedenvelope.com), in 1:1 allocation ratio. Randomization aims at equal distribution of the active treatment throughout the study period and between the different centres. To balance the groups, stratification will be conducted according to centre (Helsinki vs. Turku), developmental disability (Yes vs. No), and weight (less than 60 kg vs. 60 kg or more).

The study will be conducted in a double-blind fashion. Study treatment assignment will be blinded for both the investigators and the subject. At each local investigation site, a defined group of trained, unblinded personnel will be responsible for preparing the intravenous study drug and for delivering the drug to blinded personnel involved in the subsequent patient treatment and care. The person preparing the drug will not participate in other aspects of the study.

The blind can be broken in case a significant medical adverse event occurs (such as suspected allergic reaction). Any intentional or unintentional breaking of the blind will be recorded and reported to the sponsor as soon as possible.

Blinding and coding lists saved are managed in secure database and under the responsibility of the Chief Investigator, who has access to this database. In case of unblinding is needed, the unblinding process is conducted as follows:

Criteria for Unblinding:

Unblinding will be performed only if it is deemed essential for the immediate clinical management of a participant.

Unblinding may be initiated if a serious adverse event (SAE) occurs that, in the investigator's judgment, requires knowledge of the treatment assignment to make critical decisions for patient care.

Procedure for Unblinding:

The investigator should first attempt to contact the trial's chief investigator or research coordinator to discuss the need for unblinding. If the chief investigator or research coordinator agrees that unblinding is necessary, the randomization code will be accessed. If the chief investigator or research coordinator cannot be reached in a reasonable time frame, the investigator may proceed to unblind, documenting the reason and the time.

Accessing the Randomization Code:

The randomization code is securely stored in a sealed envelope at the trial site in patient folder and in an electronic randomization system accessible only by authorized personnel.

The investigator or treating physician must log the details of the unblinding event, including the date, time, and rationale for unblinding, in the participant's medical record, from where it transferred eCRF.

Surgery Surgery - Posterior surgery for scoliosis will be conducted according to current standard. Surgical planning of implant placement and the need for Ponte procedures will be carried out preoperatively. Each patient will be placed in the prone position and the posterior elements will be exposed using electrocautery. Ponte osteotomy will be conducted as described previously (Ponte et al, 1985). After full facetectomies, ligamentum flavum and laminae are resected for 5 mm posteriorly at three adjacent levels. The deformity will be corrected using bilateral segmental pedicle screw instrumentation and by en bloc vertebral column derotation. Spinal fusion is carried out using autograft acquired from facetectomies and osteotomies with bone graft extenders (iFactor, Cerapedics, Ic., Westminster, CO). Spinal cord monitoring (MEP, SSEP, lumbar nerve root EMG with or without pedicle screw stimulation) will be undertaken in all patients. A single subfascial drain (Hemovac Ch14; Zimmer, Warsaw, Indiana) will be placed and kept for 24 hours post-operatively. A sterile wound dressing will be applied at the end of surgery. All patients will be mobilized using a standardized protocol: sitting on the day of surgery, minimum four steps on 1st postoperative day (AIS), and progressively increasing walking distance with an aim to discharge patients on 4th -5th postoperative day. Discharge criteria include ability to walk independently (AIS) or sit independently (NMS), no need for opioid prescription, and ability to empty bladder spontaneously without a significant urinary retention (>200 mL).

Anaesthesia All patients will have total intravenous anaesthesia including dexmedetomidine, propofol and remifentanil-infusions. Mean arterial pressure will be kept between 65 mmHg and 75 mmHg during surgery and for the first 24 hours postoperatively. Cefuroxime and Vancomycin will be used as antibiotic prophylaxis. All patients will receive pain control by oral long-acting Targiniq™ twice daily along with on demand short-acting oral oxycodone. The analgesic management also includes regular oral paracetamol. All patients will receive an intravenous bolus of tranexamic acid (30 mg/kg, maximum dose 1500 mg) within 30 minutes before incision and then an infusion (10 mg/kg/h, maximum dose 500 mg/h) during surgery. Intraoperative blood loss will be measured and recorded as the amount of blood collected in the cell saver, surgical wound dressings will be weighed during surgery, excluding any irrigation with saline. Allogenic red blood cells will be transfused according to a threshold level of Hb 80 g/L during surgery or during the hospital stay. Pooled frozen human plasma will be given according to randomization or if the blood loss exceeds 50% of the patient's total blood volume (safety criteria). Platelets will be infused if the blood loss is more than 100% of the blood volume. The estimated blood volume will be calculated using a formula of 70 ml/kg x weight (kg). Arterial gas analyses will be performed minimum twice intraoperatively and at the postoperative recovery unit to rule out hyponatremia and hyperkalemia. Vasopresssin is not part of our standardized anaesthesia protocol.

Assessment Day 1 of the trial is day of the surgery, and the trial medication and placebo will be given to patients. During surgery Intraoperative blood loss is determined by weighting of surgical folds and measurement of surgical suction collection.

Mean arterial pressure (MAP), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), heart rate, blood oxygen saturation, BIS/SQI, body temperature and noradrenalin infusion (μg/kg/min) is recorded at anaesthesia induction, after patient positioning in prone position on operating table, after surgical incision, after implantation of screws and rods, after correction of scoliosis and after wound closure.

Patient haemoglobin concentration and haematocrit is recorded at end of surgery, 4 hours, and 8 hours after surgery. Pain visual analogue scale (VAS 0-10) is recorded at 4 and 8 hours after end of surgery.

Day 2 to 5 are the 1st to 3rd postoperative days. Patients are hospitalised at surgical ward. At day 2 to 5 patient haemoglobin concentration and hematocrit is recorded. At day 2 wound drain is removed and total drain output is recorded.

PCA pump is removed at day 3 and total oxycodone consumption is recorded. Peroral oxycodone consumption is recorded at day 4 to 5.

Pain VAS is recorded at day 2 to 4. Nausea, skin rash and other possible other adverse reactions are recorded.

Scoliosis radiographs, SRS-24 questionnaire, Pain VAS, adverse events, and pain medication are recorded at 6 and 24 months.

End of Trial Trial ends 24 months after surgery of the last participant. The Sponsor and/or the trial steering committee have the right at any time to terminate the study for clinical or administrative reasons.

The end-of-trial is the date of the last visit of the last subject. The end of study visit includes assessment of primary and secondary outcome measures, assessments of safety and compliance with study treatments, and recording of concomitant medications.

Unblinded interim analysis will be conducted after enrollment of 50% of the predetermined number of patients. If the experimental group shows >20% higher intraoperative blood loss, >20% higher incidence of blood transfusions or >20% higher complication rate, as compared to comparator the trial will be terminated. The analysis and possible recommendation of study termination will be made by independent external DSMB.

Description of treatment OCTAPLAS is a solvent/detergent (S/D) treated, pooled human plasma indicated for replacement of multiple coagulation factors in patients with acquired deficiencies due to liver disease or who are undergoing cardiac surgery or liver transplantation; and plasma exchange in patients with thrombotic thrombocytopenic purpura (TTP). OCTAPLAS is infused based on ABO-blood group compatibility.

OCTAPLAS is marketed in the Member States of the Union. The marketing authorisations include major surgery.

10 ml/kg OCTAPLAS (maximal dose 400 ml) is infused in 60-minute infusion prior to surgical infusion. This should increase the patient's plasma coagulation factor levels by approximately 15-25%, resulting in lower intraoperative blood loss.

PLASMALYTE Injection is a sterile, nonpyrogenic intravenous solution which does not contain bacteriostatic or antimicrobial agents or added buffers. 19 PLASMALYTE Injection pH 7.4 (Multiple Electrolytes Injection, Type 1, USP) administered intravenously has value as a source of water, electrolytes, and calories. One litre has an ionic concentration of 140 mEq sodium, 5 mEq potassium, 3 mEq magnesium, 98 mEq chloride, 27 mEq acetate, and 23 mEq gluconate. The osmolarity is 294 mOsmol/L (calc). Normal physiologic osmolarity range is 280 to 310 mOsmol/L. The caloric content is 21 kcal/L.

PLASMALYTE is marketed in the Member States of the European Union. The marketing authorisations include major surgery.

10 ml/kg (maximal dose 400 ml) PLASMALYTE is infused in 60-minute infusion prior to surgical infusion. PLASMALYTE A serves as placebo. PLASMALYTE is the standard crystalloid used in the participating investigation sites.

The study medication will be supplied to pharmacy by Helsinki and Turku University hospitals and retrieved at the end of the study. The investigator is responsible for the control of the treatments under investigation. Adequate records for the receipt and disposition of the IMP will be maintained.

The investigator will use a standard prescription manner of the institution and the research nurse will collect the medication from the pharmacy.

Accountability and subject compliance with study treatments will be assessed by maintaining dispensing and return records.

Safety reporting Adverse events will be reported according to Common Terminology Criteria for adverse effects (CTCAE, V.5, 2017) and graded as an assessment of the causal relationship to the investigational medicinal product. The PI or a delegated physician is responsible for registering and reporting AE/AR or serious AEs or serious ARs (SAE/SAR). All assessments will be documented in HUSeCRF and registered at the in-hospital treatment daily and follow-up visit at 3 months and 24 months post-surgery. Thereafter, the safety registration and reporting will be finalised. A SAE/SAR will be reported to the chief investigator within 24 hours after the PI becomes aware of event. If the PI at one of the participating sites suspects a suspected unexpected serious adverse reaction, they will inform the chief investigator with 24 hours. SUSARs will be reported to Fimea with CIOMS form, which transfers them to EudraVigilance database. If the event is fatal or life threatening, the event will be reported immediately. Any event that is neither fatal nor life threatening is reported within 7 days of the investigators' knowledge of such an event. In the case of a event, all participating investigators will be informed of the event, and any consequences related to the execution of the trial will be communicated.

Data Safety Monitoring Board The investigators and institutions involved in this clinical trial are under clinical trial-related safety monitoring. Independent Data Safety Monitoring Board (DSMB) evaluates risks and if necessary the efficacy of investigational product. DSMB recommends the sponsor either to continue or terminate the ongoing investigation. The DSMB is composed of paediatric orthopaedic surgeon, paediatrician, paediatric anaesthesiologist and biostatistician, all members of DSMB are experienced in clinical research involving underage patients. All trial documents are available to the public at the European Medicines Agency website Clinical Trials Information System (CTIS) database. If protocol deviations occur, these are reported from PIs to the chief investigator as soon as possible and noted in the eCRF separately.

Statistics The sample size has been evaluated with significance level (alpha) 5%, power (1-beta) 70% with expected mean blood loss in Plasmalyte group (NMS 1085 ml (SD 1049), AIS 554 ml (SD 349) and Octaplas (NMS 700ml, AIS 409). Expected blood loss is derived from institutional treatment registry (Soini et al NASSJ 2022). Allowing 5% lost to follow-up 97 patients for both groups are required. The statistical analyses are adjusted using linear mixed model with developmental disability diagnosis and weight as independent variables.

Intention to treat analysis set is used for primary and secondary outcomes and safety analysis set for AEs.

Data handling Data are collected locally and reported continuously after every visit to an electronic Case Report Form (HUSeCRF). The PIs at each investigative site are responsible for data entry into the HUSeCRF and for the validity of the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Aged between 10 and 21 years of age
* Scoliosis requiring posterior scoliosis surgery using all pedicle screw technique for AIS (>45-degree major curve) or NMS (>50-degree major curve)
* Normal whole spine MRI except for the spinal deformity (only for patients with adolescent idiopathic scoliosis as patients with neuromuscular scoliosis do not typically undergo MR images as they would need general anaesthesia)

Exclusion Criteria:

* Immunoglobulin A-deficiency
* Need for anteroposterior surgery
* Need for three column vertebral resection
* Smoking
* Diabetes mellitus
* Abnormalities in blood coagulation (thromboplastin time below above or below of normal values, 70-130%)
* Blood trombosytes less than 150 x E9/l
* Body mass index over 40
* Allergy or hypersensitivity to study medications or their ingredients
* Pregnancy or breast-feeding, aim of becoming pregnant during the study.
* Participation in another study and receipt of any other investigational agent during 2 year period of current investigation
* Inability to provide written informed consent
* Any significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk by participation in the study, or may influence the result of the study.
* A history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Known history of, or documented positive hepatitis B or C or HIV infection Prior or concurrent malignancy
* Aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 3 x upper-limit of normal
* Creatinine clearance (CrCl) < 60 ml/min measured by 24-hour urine collection or estimated from the Cockcroft and Gault formula
* Clinically significant ECG findings as judged by the investigator
* Amiodarone medication
* Hyperkalemia
* Renal insufficiency
* AV-block
* Metabolic or respiratory alkalosis
* Hypochlorhydria
* Hypersensitivity for active component or additives.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Exposure to closure
  Bleeding during surgery (milliliters, mL). Typical intraoperative blood loss ranges 500 mL to 3000 mL representing 20% to 75% blood loss out of total blood volume. Higher blood loss during surgery is associated with worse outcomes.

SECONDARY OUTCOMES:
Total blood loss | From exposure to drain removal at 24 hours postoperatively
  Intraoperative and drain output calculated together in milliliters (mL). Mean 24 hour drain output typically equals to intraoperative blood loss with a range from 500 mL to 1500 mL. Higher blood loss during perioperative management is associated with worse outcomes.
Need for allogeneic blood transfusion | From surgical exposure to 72 hours postoperatively
  Number of red blood cell packages infused during and after surgery until 3rd postoperative day. Use of allogeneic blood transfusion is associated with increased risk for surgical site infection and transfusion related reaction.
Health-related quality of life | At 6 and 24 months
  SRS-24 outcome questionnaire total score with 5.0 representing excellent and 1.0 the worse possible scoliosis specific health-related quality of life.
Adverse events | From surgery to 2-year follow-up
  Deep surgical site infection, skin reaction, transfusion related reaction, neurologic injury. Surgical site infection has an incidence of less than 2.0% after spinal fusion surgery and is associated with significant treatment related burden, including revision surgery and prolonged antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Ahonen, MD, Ass Prof, Ortho surgeon, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No
Sensitive clinical data. However, data will be provided upon a reasonable request to the Principal Investigator.

REFERENCES:
- [Background] Javaherforoosh Zadeh F, Janatmakan F, Shafaee Tonekaboni M, Soltanzadeh M. The Effect of Fibrinogen on Blood Loss After Lumbar Surgery: A Double-Blind Randomized Clinical Trial. Anesth Pain Med. 2019 Jun 1;9(3):e91199. doi: 10.5812/aapm.91199. eCollection 2019 Jun. PMID 31497522
- [Background] Goobie SM, Zurakowski D, Glotzbecker MP, McCann ME, Hedequist D, Brustowicz RM, Sethna NF, Karlin LI, Emans JB, Hresko MT. Tranexamic Acid Is Efficacious at Decreasing the Rate of Blood Loss in Adolescent Scoliosis Surgery: A Randomized Placebo-Controlled Trial. J Bone Joint Surg Am. 2018 Dec 5;100(23):2024-2032. doi: 10.2106/JBJS.18.00314. PMID 30516625
- [Background] Helenius I, Keskinen H, Syvanen J, Lukkarinen H, Mattila M, Valipakka J, Pajulo O. Gelatine matrix with human thrombin decreases blood loss in adolescents undergoing posterior spinal fusion for idiopathic scoliosis: a multicentre, randomised clinical trial. Bone Joint J. 2016 Mar;98-B(3):395-401. doi: 10.1302/0301-620X.98B3.36344. PMID 26920966
- [Background] Helenius L, Diarbakerli E, Grauers A, Lastikka M, Oksanen H, Pajulo O, Loyttyniemi E, Manner T, Gerdhem P, Helenius I. Back Pain and Quality of Life After Surgical Treatment for Adolescent Idiopathic Scoliosis at 5-Year Follow-up: Comparison with Healthy Controls and Patients with Untreated Idiopathic Scoliosis. J Bone Joint Surg Am. 2019 Aug 21;101(16):1460-1466. doi: 10.2106/JBJS.18.01370. PMID 31436653
- [Background] Helenius L, Gerdhem P, Ahonen M, Syvanen J, Jalkanen J, Charalampidis A, Nietosvaara Y, Helenius I. Postoperative outcomes of pedicle screw instrumentation for adolescent idiopathic scoliosis with and without a subfascial wound drain: a multicentre randomized controlled trial. Bone Joint J. 2022 Sep;104-B(9):1067-1072. doi: 10.1302/0301-620X.104B9.BJJ-2022-0391.R1. PMID 36047026
- [Background] Soini V, Raitio A, Helenius I, Helenius L, Syvanen J. A retrospective cohort study of bleeding characteristics and hidden blood loss after segmental pedicle screw instrumentation in neuromuscular scoliosis as compared with adolescent idiopathic scoliosis. N Am Spine Soc J. 2022 Dec 5;12:100190. doi: 10.1016/j.xnsj.2022.100190. eCollection 2022 Dec. PMID 36561891
- [Background] Ahonen M, Helenius I, Gissler M, Jeglinsky-Kankainen I. Mortality and Causes of Death in Children With Cerebral Palsy With Scoliosis Treated With and Without Surgery. Neurology. 2023 Oct 31;101(18):e1787-e1792. doi: 10.1212/WNL.0000000000207796. Epub 2023 Sep 7. PMID 37679048